CLINICAL TRIAL: NCT04096560
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Rising Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAK-994 in Patients With Narcolepsy With or Without Cataplexy (Narcolepsy Type 1 or Narcolepsy Type 2)
Brief Title: A Study of TAK-994 in Adults With Type 1 and Type 2 Narcolepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A safety signal has emerged in Phase 2 studies of TAK-994. As an immediate precautionary measure, Takeda has suspended dosing of patients and has decided to stop Phase 2 studies early.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-994-1501; JapicCTI-205178 (Registry Identifier: JapicCTI); 2020-000777-24 (Registry Identifier: EudraCT); U1111-1240-0346 (Registry Identifier: WHO)
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Narcolepsy Type 1 (NT1); Narcolepsy Type 2 (NT2)
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: Placebo (Placebo Comparator): TAK-994 placebo-matching tablets, orally, twice daily (BID) for 28 days, in participants with NT1.
  Interventions: Drug: Placebo
- Part A: TAK-994 120 mg (Experimental): TAK-994 120 mg, orally, BID for 28 days, in participants with NT1.
  Interventions: Drug: TAK-994
- Part A: TAK-994 180 mg (Experimental): TAK-994 180 mg, orally, BID for 28 days, in participants with NT1.
  Interventions: Drug: TAK-994
- Part B: Placebo (Placebo Comparator): TAK-994 placebo-matching tablets, orally, BID for 56 days, in participants with NT1.
  Interventions: Drug: Placebo
- Part B: TAK-994 30 mg (Experimental): TAK-994 30 mg tablets, orally, BID for 56 days, in participants with NT1.
  Interventions: Drug: TAK-994
- Part B: TAK-994 90 mg (Experimental): TAK-994 90 mg tablets, orally, BID for 56 days, in participants with NT1.
  Interventions: Drug: TAK-994
- Part B: TAK-994 180 mg (Experimental): TAK-994 180 mg tablets, orally, BID for 56 days, in participants with NT1.
  Interventions: Drug: TAK-994
- Part C: TAK-994 180 mg (Experimental): TAK-994 180 mg tablets, orally, BID for 56 days, in Chinese participants with NT1.
  Interventions: Drug: TAK-994

INTERVENTIONS:
Drug: TAK-994 — TAK-994 tablets.
  Other Names: Firazorexton
  Arms: Part A: TAK-994 120 mg; Part A: TAK-994 180 mg; Part B: TAK-994 180 mg; Part B: TAK-994 30 mg; Part B: TAK-994 90 mg; Part C: TAK-994 180 mg
Drug: Placebo — TAK-994 placebo-matching tablets.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The main aims of the study are:

* To check for side effects from TAK-994 and check what dose of TAK-994 participants can tolerate.
* To check what dose range provides adequate relief of narcolepsy symptoms.
* To check how much TAK-994 stays in the blood of participants, over time.

The study will have 4 parts. Participants can only join 1 of the parts.

A. Participants with type 1 narcolepsy will take either TAK-994 or placebo tablets for 28 days. A placebo looks just like TAK-994 but will not have any medicine in it.

B. Participants with type 1 narcolepsy will take 1 of 3 doses of TAK-994 or placebo tablets for 56 days.

C. Participants with type 1 narcolepsy in China only will take TAK-994 or placebo tablets for 56 days.

D. Participants with type 2 narcolepsy will take either TAK-994 or placebo tablets for 28 days.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-994. TAK-994 is being tested in participants with NT1 and NT2.

The study will enroll up to approximately 202 participants. The study has 4 Parts: Parts A, B, C (China only) and D. Part A - Part A has 2 cohorts [Cohorts (A1a and A1b) A2] In both of these Cohorts, participants will be randomly assigned (by chance, like flipping a coin) in a 2:1 ratio to receive TAK-994 or placebo up to 28 days:

* Part B: In Part B, participants will be randomized in 1:1:1:1 ratio in four parallel arms to receive TAK-994 Dose 1, 2 or 3 or placebo for 56 days. Depending upon their eligibility participants completing Part B of the study treatment will be enrolled to participate in an Extension study.
* Part C: In Part C, participants only from China will be enrolled and randomized in a 2:1 ratio to receive TAK-994 and placebo for 56 days.
* Part D: Participants will be included in two cohorts [Cohorts (D1a and D1b) and D2] and will be randomized in 2:1 ratio to receive TAK-994 or placebo for 28 days. The dose will be selected based on the safety and tolerability in Part A.

This multi-center trial will be conducted in the United States, Japan, China, Italy, France, and European Union. The overall duration of the study is 63 days. Participants will be followed up for 7 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of narcolepsy type 1 (NT1) (Parts A-C) or NT2 (Part D) by polysomnography (PSG)/ multiple sleep latency test (MSLT) performed within the past 10 years meeting the minimal acceptable criteria for the proper performance of the PSG/MSLT as outlined by the International Classification of Sleep Disorders, 3rd edition criteria.
2. The participant's Epworth Sleepiness Scale (ESS) score must be greater than or equal to (>=) 10 at Day -1.
3. Must be willing to discontinue all medications used for the treatment of NT1/NT2.
4. The human leukocyte antigen (HLA) genotype: Part A: should test positive for human leukocyte antigen (HLADQB1)* 06:02 (PARTs A-C)- (positive results for either homozygous or heterozygous alleles will be considered "positive" and acceptable). However, if the HLA test is negative (i.e. negative for the heterozygous allele) and the PI feels strongly that the participant has narcolepsy with cataplexy (NT1) then a discussion should be initiated between the PI and the sponsor or designee about the advisability of doing a spinal tap to determine the participant's cerebrospinal fluid (CSF) orexin-1 (OX-1) level. If the CSF result shows the orexin 1 (OX-1) concentration is either less than or equal to<110 pg/mL, or less than one-third of mean values obtained in normal participants with the same standardized assay, then the diagnosis of NT1 is established allowing the participant to be enrolled and randomized, If the CSF OX-1 concentration is >110 pg/mL then the participant will not be allowed to continue in the study .
5. For Parts A, B, and C, during the screening period, participant, must have >=4 partial or complete episodes of cataplexy/week (WCR), and >=4 partial or complete episodes of cataplexy/week during the screening period when off of anticataplexy medications, averaged over 2 weeks (14 consecutive days) minimum. WCR recording taken during following period will be considered for study eligibility: after the participant has stopped taking anticataplexy medications for at least 7 days (minimum 7-day washout) and study Day -2.

Exclusion Criteria:

1. Has a risk of suicide according to endorsement of Item 4 or 5 of the screening/baseline visit Columbia suicide severity rating scale (C-SSRS) or has made a suicide attempt in the previous 12 months.
2. Is an excessive (>600 mg/day) caffeine user 1 week before to the study screening.
3. Has a history of cancer (except carcinoma in situ that has been resolved without further treatment or basal cell skin cancer); past or current epilepsy, seizure; a lifetime history of major psychiatric disorder other than depression or anxiety; a clinically significant history of head injury or head trauma; a history of cerebral ischemia, transient ischemic attack, intracranial aneurysm, or arteriovenous malformation; known coronary artery disease, a history of myocardial infarction, angina, cardiac rhythm abnormality, or heart failure; or current or recent (within 6 months) gastrointestinal disease expected to influence the absorption of drugs. Any history of Roux-en-Y gastric bypass is considered exclusionary and any other surgical intervention that may influence the absorption of drugs should be discussed and approved by the sponsor or designee before enrolling the participants.
4. Has a medical disorder, other than narcolepsy, associated with EDS. This includes clinically significant moderate to severe obstructive sleep apnea and/or with or without treatment with mandibular advanced device hypoglossal nerve stimulation and/or positive airway pressure (PAP) therapy) and/or restless legs syndrome (RLS)/periodic limb movement disorder that has a significant impact on daytime sleepiness. This is evidenced by a clinical history of sleep apnea syndrome (loud snoring with observed respiratory pauses in the absence of nPSG) and/or RLS causing historical sleep onset/maintenance insomnia with resultant insufficient sleep. Or any as evaluated during the clinical interview at screening. pPast PSG data demonstrating any of the following sleep disturbances: apnea Hypopnea Index ≥15 or apnea index ≥10, an oxygen saturation of <80 for >10 seconds, periodic leg movement arousal index of ≥15/h) or as evaluated on interview at the time of screening. Asshould be considered exclusionary unless, based on a clinical evaluation by the investigator, a meaningful change in clinical status has occurred that would impact the results. Because nPSG data is obtained on Day -2, subjects may fail screening if criteria are not meet on the Day -2 nPSG.
5. Has a usual bedtime later than 2400 (12:00 AM, midnight) or an occupation requiring nighttime shift work or variable shift work within the past 6 months or travel within more than 3 time zones, within 14 days before Study Day -2.
6. Has a nicotine dependence that is likely to have an effect on sleep (e.g., a participant who routinely awakens at night to smoke) and/or an unwillingness to discontinue all smoking and nicotine use during the confinement portions of the study. Participants undergoing optional CSF collection.
7. Has a local infection at the puncture site.
8. Has developed signs of lumbar radiculopathy, including lower extremity pain and paresthesia.
9. Has any known focal neurological deficit that might suggest an increase in intracranial pressure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (78):
- United States (36):
  - Wright Clinical Research, Alabaster, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - CITrials - Bellflower, Bellflower, California
  - Santa Monica Clinical Trials, Los Angeles, California
  - Stanford School of Medicine, Redwood City, California
  - Pacific Research Network, Inc, San Diego, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Delta Waves Sleep Disorders and Research Center, Colorado Springs, Colorado
  - St. Francis Medical Institute, Clearwater, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - Clinical Trials of Florida, Miami, Florida
  - JSV Clinical Research Study, Inc, Tampa, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Sleep Practitioners, LLC, Macon, Georgia
  - Global Research Associates, Stockbridge, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Lutheran Sleep Disorder Center, Fort Wayne, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Helene A. Emsellem, MD PC trading as "The Center for Sleep & Wake Disorders", Chevy Chase, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Neurocare, Inc., dba Neurocare Center for Research, Newton, Massachusetts
  - Research Carolina Elite LLC, Denver, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sleep Medicine and Neuroscience Institute, Dublin, Ohio
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
- Canada (3):
  - West Ottawa Sleep Centre, Ottawa, Ontario
  - Toronto Sleep Institute, Toronto, Ontario
  - Jodha Tishon Inc., Toronto, Ontario
- China (4):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Jinan University, Tianhe, Guangdong
  - The First Hospital of Jilin University, Changchun, Jilin
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- Finland (2):
  - Terveystalo Helsinki Uniklinikka, Helsinki
  - Turku University Hospital, Turku
- France (2):
  - Hopital Gui de Chauliac, Montpellier, Herault
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
- SomnoCenter Budapest, Budapest, Hungary
- Italy (4):
  - IRCCS Oasi Maria SS, Troina, Enna
  - Universita di Bologna-Clinica Neurologica-Dipartimento di Scienze Neurologiche, Bologna
  - Ospedale San Raffaele (San Raffaele Turro), Milan
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
- Japan (15):
  - SOUSEIKAI PS Clinic, Fukuoka, Fukuoka
  - You Ariyoshi Sleep Clinic, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Kaiseikai Kita Shin Yokohama Internal Medicine Clinic, Yokohama, Kanagawa
  - Howakai Kuwamizu Hospital, Kumamoto, Kumamoto
  - Jinyukai Kotorii Isahaya Hospital, Isahaya-shi, Nagasaki
  - Shunkaikai Inoue Hospital, Nagasaki, Nagasaki
  - Gokeikai Osaka Kaisei Hospital, Osaka, Osaka
  - Kyowakai Hannan Hospital, Sakai-shi, Osaka
  - Koishikawa Tokyo Hospital, Bunkyō City, Tokyo-To
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo-To
  - Yoyogi Sleep Disorder Center, Shibuya-ku, Tokyo-To
  - Sleep Support Clinic, Shinagawa-ku, Tokyo-To
  - Sleep & Stress Clinic, Shinagawa-ku, Tokyo-To
  - Sumida Hospital, Sumida-ku, Tokyo-To
- Netherlands (2):
  - Stichting Epilepsie Instelling Nederland, Heemstede, Heemstede
  - Kempenhaeghe, Heeze, Heeze
- South Korea (2):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Hospital, Daegu
- Spain (4):
  - Hospital Universitario Araba Sede Santiago, Vitoria-Gasteiz, Alava
  - Hospital General de Castellon, Castellon, Castellon
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Vithas Nuestra Senora de America, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Dauvilliers Y, Mignot E, Del Rio Villegas R, Du Y, Hanson E, Inoue Y, Kadali H, Koundourakis E, Meyer S, Rogers R, Scammell TE, Sheikh SI, Swick T, Szakacs Z, von Rosenstiel P, Wu J, Zeitz H, Murthy NV, Plazzi G, von Hehn C. Oral Orexin Receptor 2 Agonist in Narcolepsy Type 1. N Engl J Med. 2023 Jul 27;389(4):309-321. doi: 10.1056/NEJMoa2301940. PMID 37494485
- See also: : To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a34e

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 35 investigative sites in Canada, China, France, Hungary, Italy, Japan, South Korea, Spain and United States from 27 May 2020 to 05 November 2021. The study was early terminated due to a safety signal that had emerged in the phase 2 studies of firazorexton.
Pre-assignment Details: Participants with Narcolepsy Type 1 or Type 2 were planned to be enrolled in study in Parts A, B, C and D to receive TAK-994 or placebo. Due to the early termination of the study, data was not collected for Part C: placebo and was insufficient for Part C: TAK-994 180 mg to allow the pre-planned analyses. Similarly, for Part D, the prespecified sample size at Week 4 was not reached and therefore the pre-planned analyses cannot be adequately interpreted.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Started | 7 | 7 | 8 | 17 | 17 | 20 | 19 | 2
Completed | 6 | 7 | 8 | 12 | 10 | 12 | 9 | 0
Not Completed | 1 | 0 | 0 | 5 | 7 | 8 | 10 | 2
Not completed — Reason not Specified | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Pretreatment Event, Serious Adverse Event, or Adverse Event | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 5 | 6 | 4 | 6 | 1
Not completed — Met the Discontinuation Criteria of the Protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Part A: Placebo: TAK-994 placebo-matching tablets, orally, BID for 28 days, in participants with NT1.
- Part A: TAK-994 180 mg: TAK-994 120 mg, orally, BID for 28 days, in participants with NT1
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg | Total
Number analyzed (Participants) | 7 | 7 | 8 | 17 | 17 | 20 | 19 | 2 | 97
Age, Continuous [Mean (Full Range); unit: years] | 31.4 [22 to 36] | 38.0 [23 to 53] | 33.4 [18 to 45] | 32.6 [18 to 47] | 33.4 [18 to 55] | 28.8 [18 to 48] | 29.2 [19 to 43] | 38.5 [25 to 52] | 33.16 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 8 | 12 | 10 | 12 | 1 | 54
  Male | 3 | 5 | 3 | 9 | 5 | 10 | 7 | 1 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 7 | 7 | 8 | 17 | 14 | 19 | 18 | 2 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 4 | 1 | 6 | 6 | 3 | 2 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 3 | 1 | 4 | 0 | 0 | 12
  White | 5 | 3 | 3 | 11 | 7 | 8 | 15 | 0 | 52
  More than one race | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 7
Height [Mean (Full Range); unit: centimeters (cm)] | 168.07 [157.5 to 177.8] | 176.61 [162.0 to 187.9] | 164.01 [152.8 to 177.8] | 171.00 [150.4 to 187.0] | 164.24 [151.0 to 177.8] | 168.38 [151.9 to 182.0] | 171.66 [160.0 to 185.4] | 169 [163.0 to 175.0] | 169.12 [150.4 to 187.9]
Weight [Mean (Full Range); unit: kilograms (kg)] | 85.77 [74.2 to 92.7] | 80.07 [56.7 to 102.5] | 74.33 [60.0 to 91.9] | 80.75 [46.3 to 126.5] | 71.97 [48.0 to 108.0] | 77.68 [52.3 to 102.0] | 80.33 [56.7 to 102.0] | 77 [66.0 to 88.0] | 78.48 [46.3 to 126.5]
Body Mass Index (BMI) [Mean (Full Range); unit: kilogram per square meter (kg/m^2)] — BMI= Weight (kg)/[height(m)^2]
  kilogram per square meter (kg/m^2) | 30.529 [25.3 to 37.4] | 25.629 [20.5 to 33.2] | 27.575 [23.2 to 33.8] | 27.48 [20.5 to 38.9] | 26.56 [18.2 to 38.3] | 27.29 [19.7 to 35.3] | 27.21 [19.2 to 34.0] | 26.75 [24.8 to 28.7] | 27.37 [18.2 to 38.9]
Average Sleep Latency (MWT) [Mean (Full Range); unit: minutes] — The Maintenance of Wakefulness Test (MWT) is a validated, objective measure that evaluates a person's ability to remain awake under soporific conditions for a defined period. During each MWT session (1 session = 40 minutes), participants were instructed to sit quietly and remain awake for as long as possible. Sleep latency in each session was recorded on electroencephalography (EEG). If no sleep was observed according to these rules, then the latency was defined as 40 minutes.
  minutes | 3.30 [1.1 to 8.6] | 4.41 [0.3 to 13.4] | 2.75 [1.0 to 6.9] | 6.0 [0 to 31] | 6.1 [1 to 21] | 6.1 [0 to 19] | 4.9 [0 to 23] | 17.87 [4.5 to 40] | 6.43 [0 to 40]
Epworth Sleepiness Scale (ESS) Score [Mean (Full Range); unit: score on a scale] — The ESS is a subjective, self-administered, validated scale (scored 0 to 3) to respond to each of the 8 questions of daily life that asks them how likely they are to fall asleep in those situations. The scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range.
  score on a scale | 18.6 [13 to 21] | 17.4 [13 to 24] | 18.0 [11 to 23] | 16.6 [8 to 21] | 18.5 [12 to 23] | 17.5 [10 to 23] | 17.4 [11 to 23] | 20 [16 to 24] | 18 [8 to 24]
Weekly Cataplexy Rate (WCR) [Mean (Full Range); unit: cataplexy attacks per week] — WCR = (Total number of cataplexy over a number of non-missing diary days for a given duration/number of Non-missing diary days in that duration)*7. Population: Due to early termination of the study, no secondary efficacy data was collected and analyzed for participants in Part C: TAK-994 180 mg.
  cataplexy attacks per week
    number analyzed (Participants) | 7 | 7 | 8 | 17 | 17 | 20 | 19 | 0 | 95
    (all) | 19.9 [10 to 49] | 19.1 [5 to 41] | 12.0 [4 to 28] | 15.94 [0.0 to 50.0] | 14.98 [3.5 to 72.5] | 11.68 [4.3 to 36.5] | 15.37 [3.0 to 47.5] |  | 13.62 [0.0 to 72.5]

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE) During the Study
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: First dose of study treatment to end of study follow-up (up to Day 35) in Part A
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 7 | 7 | 8
Participants | 2 | 6 | 7

2. Primary Outcome: Part A: Number of Participants Who Meet the Markedly Abnormal Value Criteria for Safety Laboratory Tests at Least Once Postdose During the Study
Description: Standard safety laboratory values (hematology, serum chemistry, urinalysis) were collected and compared to pre-specified criteria for markedly abnormal values. Markedly abnormal values criteria: Erythrocytes(10^12/L:<0.8xlower limit of normal(LLN), >1.2xupper limit of normal(ULN); Hemoglobin grams per litre(g/L):<0.8xLLN, >1.2xULN; Hematocrit voltage/volts(V/V):<0.8xLLN, >1.2xULN; Platelets(10^9/L):<75, >600; Leukocytes(10^9/L):<0.5xLLN, >1.5xULN; Alanine Aminotransferase units/litre(U/L):>3xULN, Aspartate Aminotransferase(U/L):>3xULN; Bilirubin micromoles/litre (umol/L):>1.5xULN; Alkaline Phosphatase(U/L):>3xULN; Gamma Glutamyl Transferase(U/L):>3 x ULN; Albumin(g/L):<25; Protein Total(g/L):<0.8xLLN, >1.2xULN;Glucose millimoles/litre(mmol/L):<2.8, >19.4; Calcium(mmol/L):<1.92, >2.77; Creatinine(umol/L):>1.5xULN; Urea(mmol/L):>10.7; Sodium(mmol/L):<130, >150; Potassium(mmol/L):<3.0, >5.3. Only categories with at least one participant with event are reported.
Time Frame: First dose of study treatment to end of study follow-up (up to Day 35) in Part A
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 7 | 7 | 8
Participants
  Calcium (mmol/L): <1.92 | 0 | 1 | 0
  Sodium (mmol/L): <130 | 0 | 1 | 0
  Potassium (mmol/L): >5.3 | 1 | 0 | 0

3. Primary Outcome: Part A: Number of Participants Who Meet the Markedly Abnormal Value Criteria for Vital Sign Measurements at Least Once Postdose During the Study
Description: Vital signs (body temperature and sitting blood pressure) were collected and compared to pre-specified criteria for markedly abnormal values throughout the study. Markedly abnormal values criteria: Heart Rate (beats/min): <40, >115; Systolic Blood Pressure millimeters of mercury (mmHg): <90, ≥160, Change from Pre-Dose >20, Change from Pre-Dose >30, Time-matched Change from Baseline > 20, Time-matched Change from Baseline > 30; Diastolic Blood Pressure (mmHg): <50, ≥100, Change from Pre-Dose >20, Change from Pre-Dose >30, Time-matched Change from Baseline > 20, Time-matched Change from Baseline > 30; Respiratory Rate (breaths/min): >21; Temperature Celsius (C): >38.5. Only categories with at least one participant with event are reported.
Time Frame: First dose of study treatment to end of study follow-up (up to Day 35) in Part A
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 7 | 7 | 8
Participants
  Systolic Blood Pressure (mmHg) <90 | 2 | 0 | 0
  Systolic Blood Pressure (mmHg): Change from Pre-Dose >20 | 2 | 3 | 2
  Systolic Blood Pressure (mmHg): Change from Pre-Dose >30 | 1 | 1 | 0
  Systolic Blood Pressure (mmHg): Time-matched Change from Baseline > 20 | 4 | 7 | 6
  Systolic Blood Pressure (mmHg): Time-matched Change from Baseline > 30 | 0 | 3 | 0
  Diastolic blood pressure (mmHg): Change from Pre-Dose >20 | 1 | 3 | 0
  Diastolic blood pressure (mmHg): Time-matched Change from Baseline > 20 | 1 | 4 | 3
  Temperature (C): >38.5 | 0 | 1 | 0

4. Primary Outcome: Part A: Number of Participants Who Meet the Markedly Abnormal Value Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Postdose During the Study
Description: A 12 lead ECG was performed, the ECG values were compared to pre-specified criteria for markedly abnormal values. Markedly abnormal values criteria: ECG Mean Heart Rate (beats/min): <40, >115; PR Interval milliseconds (msec): ≤80, ≥200; corrected QT interval by Fredericia (QTcF) Interval (msec): ≤300, >500, ≥30 change from baseline and >450; QRS Duration (msec): ≤80, ≥180. Only categories with at least one participant with event are reported.
Time Frame: First dose of study treatment to end of study follow-up (up to Day 35) in Part A
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 7 | 7 | 8
Participants
  PR Interval (msec): ≥200 | 0 | 1 | 2
  QTcF Interval (msec): ≥30 change from baseline and >450 | 1 | 0 | 0
  QRS Duration (msec): ≤80 | 4 | 0 | 5

5. Primary Outcome: Parts B and C: Change From Baseline in Average Sleep Latency as Assessed by the Maintenance of Wakefulness Test (MWT)
Description: MWT: validated, objective measure that evaluates person's ability to remain awake under soporific conditions for defined period. During each MWT session (1 session=40 minutes), participants were instructed to sit quietly and remain awake for as long as possible. Sleep latency in each session was recorded on electroencephalography (EEG). If no sleep had been observed according to these rules, then latency= 40 minutes. Mixed-effect model for repeated measures (MMRM) was used for analysis. Due to early termination of the study, no post-baseline efficacy data for this outcome measure was collected and analyzed for participants in Part C: TAK-994 180 mg.
Time Frame: Baseline and Week 8 (Day 56) in Parts B and C
Population: Full Analysis Set included participants who received at least 1 dose of study drug, had baseline measure and at least 1 evaluable post-dose value. Overall number of participants analyzed is the number of participants available for analyses.
Measure: Least Squares Mean (Standard Error); unit: minutes (min)
Groups:
- Part C: TAK-994 180 mg: TAK-994 180 mg tablets, orally, BID for 56 days, in participants with NT1.
Arm/Group | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Number analyzed (Participants) | 12 | 9 | 11 | 9 | 0
minutes (min) | -2.5 (2.19) | 23.9 (2.27) | 27.4 (2.17) | 32.6 (2.25) |
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: TAK-994 30 mg; Test type: Superiority; p < 0.001, MMRM — The analysis used a linear MMRM with fixed effects for baseline (Day -1 mean values), treatment, visit, and treatment-by-visit interaction. Visit was repeated factor in the model; The unstructured covariance structure was used for the repeated statement; LS Mean Difference = 26.4, 95% CI 2-sided [20.07 to 32.73], Standard Error of Mean 3.15
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: TAK-994 90 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; The unstructured covariance structure was used for the repeated statement; LS Mean Difference = 29.9, 95% CI 2-sided [23.68 to 36.07], Standard Error of Mean 3.08
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: TAK-994 180 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; The unstructured covariance structure was used for the repeated statement; LS Mean Difference = 35.0, 95% CI 2-sided [28.73 to 41.34], Standard Error of Mean 3.14

6. Secondary Outcome: Part A: Cmax: Maximum Observed Plasma Concentration After Single Dose of TAK-994 at Day 1
Time Frame: Pre-dose and at multiple time points (up to 14 hours) post-dose at Day 1 in Part A
Population: Pharmacokinetic (PK) Analysis Set included all participants who received at least 1 dose of TAK-994 and had at least 1 measurable plasma concentration. Overall number of participants analyzed is the number of participants available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 6 | 8
nanograms per milliliter (ng/mL)
  Cmax (ng/mL); Following First (AM) Dose at Day 1 | 305.5 (68.3) | 679.1 (24.5)
  Cmax (ng/mL); Following Second (PM) Dose at Day 1 | 437.1 (46.9) | 1127 (26.4)

7. Secondary Outcome: Part A: Tmax: Time of First Occurrence of Cmax After Single Dose of TAK-994 at Day 1
Time Frame: Pre-dose and at multiple time points (Up to 14 hours) post-dose at Day 1 in Part A
Population: PK Analysis Set included all participants who received at least 1 dose of TAK-994 and had at least 1 measurable plasma concentration. Overall number of participants analyzed is the number of participants available for analyses.
Measure: Median (Full Range); unit: hours (h)
Groups:
- Part A: TAK-994 120 mg: TAK-994 120 mg tablets, orally, BID for 28 days, in participants with NT1.
- Part A: TAK-994 180 mg: TAK-994 180 mg tablets, orally, BID for 28 days, in participants with NT1.
Arm/Group | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 6 | 8
hours (h)
  Tmax (h): Following First (AM) Dose at Day 1 | 1.19 [1.00 to 5.03] | 1.00 [1.00 to 5.00]
  Tmax (h): Following Second (PM) Dose at Day 1 | 2.04 [1.02 to 4.00] | 1.75 [1.42 to 2.08]

8. Secondary Outcome: Part A: AUC(0-last): Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration After Single Dose of TAK-994 at Day 1
Time Frame: Pre-dose and at multiple time points (up to 24 hours) post-dose at Day 1 in Part A
Population: PK Analysis Set included all participants who received at least 1 dose of TAK-994 and had at least 1 measurable plasma concentration. Overall number analyzed is the number of participants with data available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 6 | 8
nanograms*hour per milliliter (ng*h/mL) | 3700 (63.0) | 8559 (26.7)

9. Secondary Outcome: Part A: Cmax: Maximum Observed Plasma Concentration After Multiple Doses of TAK-994 at Day 28
Time Frame: Pre-dose and at multiple time points (up to 14 hours) post-dose at Day 28 in Part A
Population: PK Analysis Set included all participants who received at least 1 dose of TAK-994 and had at least 1 measurable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 7 | 8
ng/mL
  Cmax (ng/mL); Following First (AM) Dose at Day 28 | 377.5 (36.6) | 856.9 (31.6)
  Cmax (ng/mL); Following Second (PM) Dose at Day 28 | 416.0 (40.9) | 829.4 (28.4)

10. Secondary Outcome: Part A: Tmax: Time of First Occurrence of Cmax After Multiple Doses of TAK-994 at Day 28
Time Frame: Pre-dose and at multiple time points (up to 14 hours) post-dose at Day 28 in Part A
Population: as for outcome 9
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 7 | 8
hours (h)
  Tmax (h): Following First (AM) Dose at Day 28 | 1.03 [0.93 to 3.10] | 1.00 [0.90 to 1.00]
  Tmax (h): Following Second (PM) Dose at Day 28 | 2.15 [2.00 to 4.05] | 3.46 [1.50 to 7.00]

11. Secondary Outcome: Part A: AUC(0-t): Area Under the Concentration-time Curve From Time 0 to Time Tau Over a Dosing Interval of TAK-994 at Day 28
Time Frame: Pre-dose and at multiple time points (Up to 12 hours) post-dose at Day 28 in Part A
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg
Number analyzed (Participants) | 7 | 8
ng*h/mL | 2968 (33.1) | 6438 (22.6)

12. Secondary Outcome: Parts B and C: Change From Baseline in the Epworth Sleepiness Scale (ESS) Total Score to Week 8
Description: The ESS is a subjective, self-administered, validated scale (scored 0 to 3) to respond to each of the 8 questions of daily life that asks participants how likely they are to fall asleep in those situations. The scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range. MMRM was used for analysis. Due to early termination of the study, no post-baseline secondary efficacy data for this outcome measure was collected and analyzed for participants in Part C: TAK-994 180 mg.
Time Frame: Baseline and Week 8 (Day 56) in Parts B and C
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Number analyzed (Participants) | 12 | 10 | 11 | 9 | 0
score on a scale | -2.1 (1.35) | -12.2 (1.41) | -13.5 (1.32) | -15.1 (1.41) |
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: TAK-994 30 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; The unstructured covariance structure was used for the repeated statement; LS Mean Difference = -10.1, 95% CI 2-sided [-14.07 to -6.16], Standard Error of Mean 1.96
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: TAK-994 90 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; The unstructured covariance structure was used for the repeated statement; LS Mean Difference = -11.4, 95% CI 2-sided [-15.20 to -7.56], Standard Error of Mean 1.89
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: TAK-994 180 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; The unstructured covariance structure was used for the repeated statement; LS Mean Difference = -13.0, 95% CI 2-sided [-16.96 to -9.09], Standard Error of Mean 1.95

13. Secondary Outcome: Parts B and C: Change From Baseline in Weekly Cataplexy Rate (WCR) at Week 8
Description: Participants will complete a daily patient-reported sleep diary to record self-reported narcolepsy symptoms. Participants will record episodes of cataplexy in the diary. The total number of events averaged for a week will be reported. WCR = (Total number of cataplexy over a number of non-missing diary days for a given duration/number of Non-missing diary days in that duration)*7. MMRM was used for the analysis. Due to early termination of the study, no secondary efficacy data was collected and analyzed for participants in Part C: TAK-994 180 mg.
Time Frame: Baseline and Week 8 (Day 56) in Parts B and C
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cataplexy attacks per week
Groups:
- Part B: TAK-994 180 mg; Part C: TAK-994 180 mg: TAK-994 90 mg tablets, orally, BID for 56 days, in participants with NT1.
Arm/Group | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Number analyzed (Participants) | 10 | 10 | 11 | 8 | 0
cataplexy attacks per week | -6.58 (7.433) | -16.17 (20.979) | -11.91 (10.174) | -15.74 (9.978) |
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: TAK-994 30 mg; Test type: Superiority; p = 0.002, MMRM — The incidence rate was the exponentiated LS means and the incidence rate ratio (IRR) was the exponentiated LS mean differences from the generalized estimating equation (GEE) Poisson regression model; The Poisson regression with natural log link was on the count of cataplexy per week; IRR = 0.05, 95% CI 2-sided [0.007 to 0.317]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: TAK-994 90 mg; Test type: Superiority; p = 0.019, MMRM — The incidence rate was the exponentiated LS means and the IRR was the exponentiated LS mean differences from the GEE Poisson regression model; The Poisson regression with natural log link was on the count of cataplexy per week; IRR = 0.20, 95% CI 2-sided [0.050 to 0.767]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: TAK-994 180 mg; Test type: Superiority; p = 0.001, MMRM — [p-value comment as in outcome 13, analysis 2]; The Poisson regression with natural log link was on the count of cataplexy per week; IRR = 0.15, 95% CI 2-sided [0.047 to 0.482]

14. Secondary Outcome: Parts B and C: Number of Participants Who Experience at Least 1 TEAE During the Study
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: First dose of study drug to end of study follow-up (up to Day 63) in Parts B and C
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: FTAK-994 90 mg: TAK-994 90 mg tablets, orally, BID for 56 days, in participants with NT1.
Arm/Group | Part B: Placebo | Part B: TAK-994 30 mg | Part B: FTAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Number analyzed (Participants) | 17 | 17 | 20 | 19 | 2
Participants | 4 | 13 | 17 | 14 | 2

15. Secondary Outcome: Parts B and C: Number of Participants Who Met the Markedly Abnormal Value Criteria for Safety Laboratory Tests at Least Once Postdose During the Study
Description: Standard safety laboratory values (serum chemistry, hematology, and urine analysis) were collected and compared to pre-specified criteria for Markedly Abnormal Values throughout the study. Markedly abnormal values criteria: Alanine Aminotransferase (U/L):>3xULN, Aspartate Aminotransferase(U/L):>3xULN; Bilirubin micromoles/litre (umol/L):>1.5xULN; Calcium(mmol/L):<1.92, >2.77; Potassium(mmol/L):<3.0, >5.3. Only categories with at least one participant with event are reported.
Time Frame: Up to Day 63 in Parts B and C
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Number analyzed (Participants) | 17 | 17 | 20 | 19 | 2
Participants
  Alanine Aminotransferase (ALT) [U/L)]: >3 × Upper limit normal (ULN) | 0 | 0 | 3 | 2 | 0
  Aspartate Aminotransferase (AST) [(U/L)]: >3 × ULN | 0 | 0 | 1 | 2 | 0
  Bilirubin (µmol/L): >1.5 × ULN | 0 | 0 | 0 | 1 | 0
  Calcium (mmol/L): <1.92 | 1 | 0 | 0 | 0 | 0
  Potassium (mmol/L): <3.0 | 1 | 0 | 0 | 0 | 0
  Potassium (mmol/L): >5.3 | 1 | 1 | 0 | 0 | 0

16. Secondary Outcome: Parts B and C: Number of Participants Who Met the Markedly Abnormal Value Criteria for Vital Sign Measurements at Least Once Postdose During the Study
Description: Vital signs (body temperature and sitting blood pressure) were collected and compared to pre-specified criteria for markedly abnormal values throughout the study. Markedly abnormal values criteria: Systolic Blood Pressure millimeters of mercury (mmHg): <90, ≥160, Change from Pre-Dose >20, Change from Pre-Dose >30, Time-matched Change from Baseline > 20, Time-matched Change from Baseline > 30; Diastolic Blood Pressure (mmHg): <50, ≥100, Change from Pre-Dose >20, Change from Pre-Dose >30, Time-matched Change from Baseline > 20, Time-matched Change from Baseline > 30; Respiratory Rate (breaths/min): >21.Only categories with at least one participant with event are reported.
Time Frame: Up to Day 63 in Parts B and C
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Number analyzed (Participants) | 17 | 17 | 20 | 19 | 2
Participants
  Systolic blood pressure (mmHg): <90 | 2 | 3 | 1 | 1 | 1
  Systolic blood pressure (mmHg):>=160 | 1 | 0 | 0 | 1 | 0
  Systolic blood pressure (mmHg): Change from Predose >20 | 5 | 7 | 10 | 10 | 0
  Systolic blood pressure (mmHg): Change from Predose >30 | 2 | 2 | 6 | 5 | 0
  Systolic blood pressure (mmHg): Time-matched Change from Baseline >20 | 2 | 11 | 13 | 14 | 1
  Systolic blood pressure (mmHg): Time-matched Change from Baseline >30 | 1 | 4 | 3 | 5 | 0
  Diastolic blood pressure (mmHg): <50 | 0 | 1 | 1 | 2 | 0
  Diastolic blood pressure (mmHg): >=100 | 1 | 1 | 2 | 2 | 1
  Diastolic blood pressure (mmHg): Change from Predose >20 | 0 | 3 | 5 | 9 | 0
  Diastolic blood pressure (mmHg): Change from Predose >30 | 0 | 0 | 1 | 3 | 0
  Diastolic blood pressure (mmHg): Time-matched Change from Baseline >20 | 2 | 5 | 7 | 7 | 0
  Diastolic blood pressure (mmHg): Time-matched Change from Baseline >30 | 0 | 0 | 1 | 2 | 0
  Respiratory Rate [Breaths per minute (breaths/min)]: >21 | 0 | 2 | 0 | 1 | 1

17. Secondary Outcome: Parts B and C: Number of Participants Who Met the Markedly Abnormal Value Criteria for ECG Parameters at Least Once Postdose During the Study
Description: A 12 lead ECG was performed, the ECG values were compared to pre-specified criteria for markedly abnormal values. Markedly abnormal values criteria: PR Interval (msec): ≤80, ≥200; QRS Duration (msec): ≤80, ≥180. Only categories with at least one participant with event are reported.
Time Frame: Up to Day 63 in Parts B and C
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
Number analyzed (Participants) | 17 | 17 | 20 | 19 | 2
Participants
  PR Interval (msec): >=200 | 2 | 2 | 1 | 3 | 0
  QRS Duration (msec):<=80 | 4 | 3 | 7 | 4 | 0

ADVERSE EVENTS:
Time Frame: First dose of study treatment to end of study follow-up (up to Day 35 in Part A and up to Day 63 in Parts B and C)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part A: Placebo | Part A: TAK-994 120 mg | Part A: TAK-994 180 mg | Part B: Placebo | Part B: TAK-994 30 mg | Part B: TAK-994 90 mg | Part B: TAK-994 180 mg | Part C: TAK-994 180 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/17 | 0/17 | 0/20 | 0/19 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/17 | 0/17 | 0/20 | 1/19 | 0/2
Other Adverse Events (participants affected / at risk) | 2/7 | 6/7 | 7/8 | 4/17 | 13/17 | 17/20 | 14/19 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=7) | Part A: TAK-994 120 mg (N=7) | Part A: TAK-994 180 mg (N=8) | Part B: Placebo (N=17) | Part B: TAK-994 30 mg (N=17) | Part B: TAK-994 90 mg (N=20) | Part B: TAK-994 180 mg (N=19) | Part C: TAK-994 180 mg (N=2)
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=7) | Part A: TAK-994 120 mg (N=7) | Part A: TAK-994 180 mg (N=8) | Part B: Placebo (N=17) | Part B: TAK-994 30 mg (N=17) | Part B: TAK-994 90 mg (N=20) | Part B: TAK-994 180 mg (N=19) | Part C: TAK-994 180 mg (N=2)
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ex-tobacco user (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glutamate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypervigilance (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 1 | 0 | 2 | 3 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 5 | 10 | 8 | 1
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 3 | 5 | 1 | 5 | 10 | 6 | 2
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Puncture site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 3 | 2 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
A safety signal had emerged in the phase 2 studies of firazorexton causing early termination of Part C and Part D of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04096560/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT04096560/SAP_001.pdf